CLINICAL TRIAL: NCT00003984
Title: Phase II Trial With a Recombinant Humanized Anti-CD33 Monoclonal Antibody (HuM195) in Patients With High Risk Primary Myelodysplastic Syndromes
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Primary Myelodysplastic Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-13981; EORTC-13981
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — lintuzumab

INTERVENTIONS:
Biological: lintuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have primary myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the therapeutic activity of monoclonal antibody HuG1-M195 on peripheral blood and bone marrow blast cell count, blood leukocyte, reticulocyte, and platelet counts, and hemoglobin levels in patients with myelodysplastic syndrome with refractory anemia with excess blasts (RAEB) (greater than 10% bone marrow myeloblasts) or RAEB in transformation. II. Assess the efficacy of this drug in terms of duration of response in these patients. III. Evaluate the toxicity of this drug in these patients.

OUTLINE: Patients receive monoclonal antibody HuG1-M195 IV over 4 hours on days 1-4. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with progressive disease after 2 courses are removed from study. Patients with stable disease receive no further treatment after 4 courses. Patients with complete or partial response receive treatment for 4 additional courses. Patients are followed at 11 and 39 days after end of course 4, monthly for 4 months, then every 3 months thereafter for 1 year from study entry.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary myelodysplastic syndrome (MDS) with greater than 10% bone marrow blasts Refractory anemia with excess blasts (RAEB) OR RAEB in transformation No chronic myelomonocytic leukemia No secondary MDS after prior chemotherapy except if treatment was for acute myeloid leukemia No allogeneic bone marrow transplantation planned

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Hemoglobin no greater than 10 g/dL OR transfusion requirement of at least 3 packs of RBCs per month OR Platelet count less than 50,000/mm3 OR Absolute neutrophil count less than 1,000/mm3 No disseminated intravascular coagulation defined as fibrinogen less than 100 mg/dL AND prolonged PT, PTT, or thrombin time AND platelet count less than 25,000/mm3 without transfusion Hepatic: Bilirubin no greater than 2.0 mg/dL Alkaline phosphatase no greater than 4 times upper limit of normal (ULN) (unless due to underlying disease or Gilbert's syndrome) SGPT and SGOT no greater than 4 times ULN (unless due to underlying disease or Gilbert's syndrome) Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No uncontrolled hypertension No congestive heart failure, cardiac arrhythmia, or angina pectoris No history of myocardial infarction within the past 6 months No other significant cardiovascular disease LVEF within normal range by MUGA or echocardiogram No active ischemia Pulmonary: No pulmonary dysfunction Other: No central or peripheral neuropathy No uncontrolled or unstable diabetes No other significant organ system dysfunction HIV negative No prior malignancy except basal cell carcinoma or carcinoma in situ of the uterus No active, uncontrolled infection Not pregnant or nursing Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 2 months since prior biologic therapy (e.g., hematopoietic growth factors or biological response modifiers) Chemotherapy: See Disease Characteristics At least 2 months since prior chemotherapy Endocrine therapy: At least 2 months since prior endocrine therapy Radiotherapy: At least 2 months since prior radiotherapy Concurrent radiotherapy allowed Surgery: At least 2 months since prior surgery Other: No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-02

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Zwierzina, MD, Study Chair — Medical University Innsbruck
Locations (27):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Ludwig Institute for Cancer Research-Brussels Branch, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Herlev Hospital - University Hospital of Copenhagen, Herlev, Denmark
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- Netherlands (5):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - C.R.C. Beatson Laboratories, Glasgow, Scotland